CLINICAL TRIAL: NCT05911334
Title: Assessing the Feasibility of the Restorative Occupational Approaches for Disordered Eating (ROADE) Program
Brief Title: Feasibility of the ROADE Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The ROADE grant was terminated early by C&G and the PI left the institution.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00006140; AOTFIRG23Hardison (Other Grant/Funding Number: American Occupational Therapy Foundation)
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Bulimia Nervosa; Anorexia Nervosa; Binge-Eating Disorder; Avoidant/Restrictive Food Intake Disorder
Keywords: Occupational Therapy; Chronic Illness Management; Eating Disorder; Yoga; Mindfulness
MeSH Terms: conditions — Bulimia Nervosa; Anorexia Nervosa; Binge-Eating Disorder; Avoidant Restrictive Food Intake Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Restorative Occupational Approaches for Disordered Eating (ROADE) (Experimental): Novel Outpatient Occupational Therapy Intervention using chronic illness management strategies, yoga, meditation for disordered eating. 8-weeks with 2 visits per week each lasting 1 hour.
  Interventions: Behavioral: ROADE Program

INTERVENTIONS:
Behavioral: ROADE Program — Outpatient Behavioral Intervention for Eating Disorder

SUMMARY:
Occupational therapy is uniquely poised to help address chronic Eating Disorders (EDs) because of our holistic approach to client care. The complex and serious nature of EDs spans so many areas of life and wellbeing, it requires an intervention strategy that addresses the whole person across mental, physical, social, and spiritual realms. Unfortunately, specialized care for EDs can be difficult to find - especially for those not sick enough to be admitted to an inpatient facility but who are still struggling to thrive in daily life. For example, in New Mexico there is only one inpatient treatment center for EDs and no specialized outpatient services. This leaves many people suffering from EDs without options for care because they are not yet sick enough. There is a need for novel interventions in this setting that go beyond the traditional weight and food-focused medical interventions and seek to help empower individuals, work around challenges, and live their lives to the fullest.

To meet this need in our community, the study team is developing a preliminary outpatient treatment program. The ROADE (Restorative Occupational Approaches for Disordered Eating) Program is an 8-week, structured, multimodal intervention seeking to reduce psychosocial symptoms and improve self-management skills for disordered eating. The intervention strategies range from: (1) wellness activities like mindfulness meditation to improve interoception, self-acceptance, and as a self-guided coping tool (2) adaptation of health management and self-care occupations to improve daily functioning while navigating ongoing disordered eating symptoms and (3) light exercise like Yoga and lymphatic drainage exercises to reconnect in a positive way with the body, improve digestion, promote relaxation, and reduce muscle tension. The current research investigates the feasibility and acceptability of this intervention while testing preliminary effects on eating disorder symptoms.

DETAILED DESCRIPTION:
Eating Disorders (ED) are pervasive, long-lasting conditions that are exceptionally destructive to wellbeing and many areas of occupational performance. In the United States an estimated 29 million individuals will suffer from an eating disorder across their lifespan (Academy for Eating Disorders, 2020) with the most common diagnoses being Anorexia Nervosa, Binge Eating Disorder, Bulimia Nervosa, and Avoidant, Restrictive, Food Intake Disorder (ARFID). Though distinct, each of these diagnoses share a feature of individuals developing a dysfunctional relationship with food that is rigid and ritualized. The point prevalence of all eating disorders combined appears to be on the rise worldwide, increasing from an estimated 4% to 8% of the population starting in the year 2000 through 2018 (Galmiche, 2019). Often this is accompanied with compulsive routines that exhaust many hours a day. Beyond disrupted eating, symptoms span almost all areas of occupation (e.g., hygiene, social functioning, work, rest) and affect both mental health and physical health (Bradford et al., 2015).

Unfortunately, with current treatments for eating disorders, the long-term outcomes are poor. Recovery can be a long process, often taking 6 years or more (Franco, 2017), but this is likely an underestimate due to the limited length of research follow up (Arcelus et al., 2011). Estimates of recovery and mortality range greatly depending on the source with as much as half of individuals not recovering fully and up to an astounding 5% of those afflicted with Anorexia Nervosa dying from the disorder (Franko et al., 2013). Sadly, 1 in 5 deaths from Anorexia Nervosa result from suicide while predictors of higher mortality include alcohol misuse and other comorbid mental health diagnoses (Arcelus et al., 2011). Multiple systematic reviews report that current interventions have yet to demonstrate strong effect sizes and there is no one specific approach that has emerged as best practice (Kotilahti et al., 2020; Murray et al., 2018; Peat et al., 2017; Zeeck et al., 2018). There is a call to move beyond a simplistic treatment model that over-emphasizes weight gain or loss and instead more fully addresses personal and social effects of the disorder, uses harm reduction strategies, and strives to empower clients (Hay et al., 2012).

The present project addresses the serious, complex, and enduring nature of eating disorders. Occupational therapy is uniquely poised to help address chronic EDs because of our holistic approach to client care. As eating disorders affect myriad areas of health and wellbeing, they require intervention strategies that addresses the whole person across mental, physical, and social realms. Specialized care for EDs can be difficult to find. This is especially true for those not sick enough to be admitted to an inpatient facility but who are still struggling to thrive in daily life. Specific to the state of New Mexico, where the project will be conducted, there are currently no outpatient mental health services that specialize in treating eating disorders. Individuals may succeed in graduating from the single in-patient eating disorder clinic in our state, but are discharged without a strong outpatient program to follow their care. This presents a large risk of relapse. Our hope is that ROADE Program will eventually grow into a resource for the community and help bridge this gap in services. More broadly, the present project has the opportunity to build a role for occupational therapists in treating eating disorders and expand our role in chronic illness management.

Occupational therapy interventions in this setting, to our knowledge, have yet been evaluated experimentally. Much of the publications in occupational therapy about eating disorder treatment is older evidence or relies on expert opinion and nonsystematic literature review to describe potential avenues for intervention (e.g. Bradford et al., 2015; Clark & Nayar, 2012; Gardener & Brown, 2010; Horner, 2006). One occupational therapy text in mental health (Crouch & Alers, 2014), one survey of occupational therapists working in mental health settings (Klockzko & Ikiugu, 2006), and a small subjective study that polled participants opinion about the helpfulness of the intervention (Biddiscombe et al., 2018) demonstrate that occupational therapy self-identifies as having a role in treating eating disorders. Key points of interest for from these perspectives are that occupational therapists should work in a collaborative model with other healthcare providers, use a holistic approach to care, and focus on the areas of occupation that are affected by the disorder. With this emerging level of evidence, the study team has developed one such program from the ground up. Our preliminary take on developing an intervention used best available evidence from within occupational therapy, but also draws from outside the profession. We focused on restorative approaches fitting within the occupational therapy practice area based on the OT Practice Framework (AOTA, 2020). This became the ROADE (Restorative Occupational Approaches for Disordered Eating) Program.

The ROADE Program is to our knowledge the first of its kind being an occupational-therapy-specific intervention for disordered eating. In its current form it is an 8-week, structured, multimodal intervention seeking to reduce psychosocial symptoms and improve self-management skills for disordered eating. The intervention strategies range from: (1) Light exercises and Yoga to improve lymphatic drainage, improve digestion, promote relaxation, and reduce muscle tension (Gibson & Mehler, 2019; Moser, 2020; Sim et al, 2017; Souza et al, 2018), (2) mindfulness meditation to improve interoception, self-acceptance, and as a self-guided coping tool (Sala et al., 2020), and (3) adaptation of health management and self-care occupations to improve daily functioning while navigating ongoing disordered eating symptoms (Crouch & Alers, 2014; Sørlie et al., 2020). It is our hope to further hone this program into a manualized intervention, track the preliminary effects of the intervention, collect feasibility data points, and then seek funding for an efficacy trial. These objectives will be explored in the form of three specific aims:

Specific Aim 1. To establish the feasibility of implementing the ROADE Program in a research setting Specific Aim 2. To determine the preliminary effects the ROADE Program intervention has on disordered eating symptoms.

Specific Aim 3. To hone the ROADE Program protocol by leveraging expert guidance, training, and experience.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Binge Eating Disorder, Anorexia Nervosa, Bulimia Nervosa, or ARFID
* Able to answer surveys in English
* 14 years of age or older

Exclusion Criteria:

* Unable to comfortably do light exercise such as Yoga

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Yale-Brown-Cornell Eating Disorder Scale | 8 weeks
  Eating Disorder Symptom Burden

SECONDARY OUTCOMES:
Beck Anxiety Inventory | 8 weeks
  Self-reported Anxiety
SF-36 | 8 weeks
  health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States